CLINICAL TRIAL: NCT06385587
Title: Technology-based Symptom Monitoring Intervention for Locally Advanced Head and Neck Cancer Patients Initiating Chemoradiation: A Pilot Study
Brief Title: Technology-based Symptom Monitoring Intervention for Locally Advanced Head and Neck Cancer Patients
Acronym: SYMTECH01
Status: Completed | Type: Observational
Sponsor: Aptar Digital Health (Industry)
Responsible Party: Sponsor
Other Study IDs: ADH-OL-Study-01-23
Record Dates: First submitted 2024-04-12; First posted 2024-04-26 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Oleena — Oleena™ is a software medical device for patients and their healthcare team which digitalizes some aspects of their supportive care, allows remote monitoring by healthcare professionals (HCP) and supports the management of targeted symptoms in adult cancer patients while they are being actively treated for their cancer.

SUMMARY:
The goal of this observational study is to assess the satisfaction and usability of an interactive and patient-centered mobile application (app), Oleena™, designed to assist head and neck cancer patients undergoing chemoradiation in managing common and distressing symptoms in real-time, as well as to assess the satisfaction and usability of the related HCP web portal. Additional secondary usage and clinical endpoints that would be used to assess intervention efficacy in future trials will be collected.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Planned to initiate chemoradiation for locally advanced head and neck cancer at Moffitt Cancer Center
* ECOG performance status ≤2
* Able to speak and read US English or Spanish
* Able to provide informed consent
* Owns a smartphone with an iOS or Android operating systemcompatible with Oleena
* Able to access the internet
* Willing to use a mobile app for symptom management

Exclusion Criteria:

* Documented or observable psychiatric or neurological disorders that would interfere with study participation (e.g., psychosis, active substance abuse).
* A prior cancer diagnosis except for non-melanoma skin cancer.
* Currently enrolled in an industry-sponsored clinical trial.
* Pregnant women.
* Patients undergoing RE-irradiation
* Patients who meet the inclusion criteria may be excluded at Investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced head and neck cancer initiating chemoradiation. Patients will use Oleena for 90 days from the initiation of the treatment and be instructed to enter symptoms as they occur and receive self-management recommendations via the app. Surveys will be completed by patients at baseline, 30, and 90 days after initiation. A subgroup of patients (20) will be asked to participate in exit interviews with a study team member regarding their experience with the app.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Users' satisfaction | End of study - Day 90 +/-10 from first radiotherapy
  Users' (participants and HCPs) level of satisfaction with the symptom management app, which will be assessed via a validated, 4-item scale, Acceptability of Intervention Measures (score range 0-20)

SECONDARY OUTCOMES:
Feasibility of the technology enabled symptom management solution | Assessed up to 90 days
  The extent to which the symptom management app can be successfully implemented within the Head and Neck Clinic. A series of objective measures (e.g., recruitment, retention, data completion, and app usage rates) will be used to define feasibility in this specific head and neck cancer population.
Usability of the technology enabled symptom management solution | Day 30 and Day 90 +/-10 from first radiotherapy
  The extent to which participants can use the symptom management app to manage their symptoms with efficiency and satisfaction and will be measured using the system usability scale (SUS) (score range 0-100)
Appropriateness of the recommendations | After 15 and then 30 patients have reached Day 30 and then Day 90
  Participating providers will rate the appropriateness of the recommendations provided by the Oleena app through a brief electronic survey
Semi-structured exit interviews | End of study - Day 90 +/-10 from first radiotherapy
  The first twenty (20) study participants exiting the study will gauge their overall perceptions regarding the intervention and identify any potential barriers and facilitators that may affect intervention implementation

OTHER OUTCOMES:
Symptom burden will be measured using the NIH PRO-CTCAE measurement system, which includes validated scales for individual toxicities | Baseline, Day 30 and Day 90 +/-10 from first radiotherapy
  The following PRO-CTCAE items will be used: diarrhea, nausea, loss of appetite, vomiting, pain, skin rash, hand-foot syndrome, fatigue, fever, breathing, cough, swallowing difficulties, mucositis, and smell and taste changes.
Quality of life will be measured using the previously validated FACT-G scale | Baseline, Day 30 and Day 90 +/-10 from first radiotherapy
  The FACT-G is a 27-item questionnaire that measures four domains of health-related quality of life including physical, social, functional, and emotional well-being with a 7-day recall period
Treatment adherence | Assessed up to 90 days
  Treatments prescribed and received, dosage, duration of treatment, dose reductions, and discontinuation
Health-economic outcome | Assessed up to 90 days
  The number of unscheduled outpatient visits, unscheduled inpatient hospitalizations and ER admissions related to the targeted symptoms
Complaints, alleged deficiencies or malfunctions of the device reported | Assessed up to 90 days
  Safety of the device

CONTACTS AND LOCATIONS:
Overall Officials: Amir Alishahi, MD, PhD, MPH, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States